CLINICAL TRIAL: NCT01570179
Title: Sugammadex in Patients Undergoing Bariatric Surgery: An Equivalence Trial Comparing Real and Ideal Body Weight-based Dosing
Brief Title: Sugammadex-dosing in Bariatric Patients
Acronym: SugReBaCh-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011-005504-14
Record Dates: First submitted 2012-03-27; First posted 2012-04-04 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Neuromuscular Blockade
Keywords: bariatric surgery; residual paralysis; surgical conditions

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- deep block ideal body weight (Experimental)
  Interventions: Drug: ideal body weight based sugammadex reversal of deep block
- deep block real body weight (Active Comparator)
  Interventions: Drug: real body weight based sugammadex reversal of deep block
- moderate block ideal body weight (Experimental)
  Interventions: Drug: ideal BW based sugammadex reversal of moderate block
- moderate block real body weight (Active Comparator)
  Interventions: Drug: real body weight based sugammadex reversal of moderate block

INTERVENTIONS:
Drug: ideal BW based sugammadex reversal of moderate block — 2 mg/kg sugammadex (based og ideal body weight)
  Arms: moderate block ideal body weight
Drug: real body weight based sugammadex reversal of moderate block — 2 mg/kg sugammadex (based on real BW)
  Arms: moderate block real body weight
Drug: real body weight based sugammadex reversal of deep block — 4 mg/kg sugammadex (based on real BW)
  Arms: deep block real body weight
Drug: ideal body weight based sugammadex reversal of deep block — 4 mg/kg sugammadex (based on ideal BW)
  Arms: deep block ideal body weight

SUMMARY:
Should the dose of sugammadex in morbid obese patients be calculated on the real body weight or the ideal body weight?

The main objective of the trial is to compare in patients undergoing bariatric surgery the efficacy of sugammadex to obtain a TOF-ratio of 100% within 3 min when dosing is based on real body weight (control intervention) with dosing based on ideal body weight (experimental intervention). The research hypothesis is that both dosing regimens are equivalent

The secondary objective of the trial is to compare the impact of the depth of neuromuscular blockade on the surgical conditions: deep block (TOF-count 1 - 3) will be compared with very deep block (TOF count = 0 and PTC < 5)

ELIGIBILITY:
Inclusion Criteria:

adult patients undergoing bariatric surgery according to the respective criteria of the French Medical Authority (HAS) and having given their written informed consent after appropriate information

Exclusion Criteria:

not fulfilling the inclusion criteria, known or suspected allergy to any of the drugs used in that study, absence of written informed consent,doubt of pregnancy in women of childbearing age, pregnancy and breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-05; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
100% TOF-recovery 3 min after sugammadex | 3 min

SECONDARY OUTCOMES:
impact of depth of block on surgical conditions | every 15 min during surgery
  to evaluate the impact of neuromuscular blockade on surgical conditions, the The "King Score" (King M, Anesthesiology 2000; 93:1392 - 7) will be applied every 15 min throught surgery by the surgeon (blinded to the study protocol)King-Score: from 1 to 4 with 1 excellent conditions, 2 good conditions, 3 acceptable conditions and 4 poor conditions.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU Strasbourg Hôpital Civil, Strasbourg, Alsace
  - CHU Nancy, Vandœuvre-lès-Nancy, Lorraine